CLINICAL TRIAL: NCT02227693
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Once-daily Oral Avatrombopag in Japanese Subjects With Chronic Liver Disease and Thrombocytopenia
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Once-daily Oral Avatrombopag in Japanese Subjects With Chronic Liver Diseases and Thrombocytopenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E5501-J081-204
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2017-12

CONDITIONS: Thrombocytopenia Associated With Chronic Liver Disease
Keywords: Thrombocytopenia; Chronic Liver Disease
MeSH Terms: conditions — Thrombocytopenia | interventions — avatrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- avatrombopag 20-mg (Experimental): 20 mg avatrombopag (1 x 20 mg tablet and 2 x 20 mg matching placebo tablets) once daily on Days 1 through 5
  Interventions: Drug: avatrombopag
- avatrombopag 40-mg (Experimental): 40 mg avatrombopag (2 x 20 mg tablets and 1 x 20 mg matching placebo tablet) once daily on Days 1 through 5
  Interventions: Drug: avatrombopag
- avatrombopag 60-mg (Experimental): 60 mg avatrombopag (3 x 20 mg tablets) once daily on Days 1 through 5
  Interventions: Drug: avatrombopag
- placebo l (Placebo Comparator): Placebo (3 x 20-mg matching placebo tablets) once daily on Days 1 through 5
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: avatrombopag — E5501 (avatrombopag) 20-mg tablets
  Arms: avatrombopag 20-mg; avatrombopag 40-mg; avatrombopag 60-mg
Drug: Placebo — Placebo matching 20-mg tablets
  Arms: placebo l

SUMMARY:
This is a phase 2, randomized, double-blind, placebo-controlled, parallel group study using avatrombopag for Japanese subjects with thrombocytopenia associated with chronic liver disease. This study will assess the effect of avatrombopag on platelet counts in Japanese subjects. Subjects will be enrolled into 2 cohorts according to the mean platelet count measured at Screening and Baseline. Within the lower baseline platelet count cohort (less than 40 x 10^9/L), subjects will be randomized in a 1:1:1:3 ratio to receive placebo, 20 mg avatrombopag, 40 mg avatrombopag, or 60 mg avatrombopag for 5 days. Within the higher baseline platelet count cohort (from 40 to less than 50 x 10^9/L), subjects will be randomized in a 2:1:2 ratio to receive placebo, 20 mg avatrombopag, or 40 mg avatrombopag for 5 days.

DETAILED DESCRIPTION:
This study will consist of Prerandomization Phase and Randomization Phase. The Prerandomization Phase includes a Screening Period (Day -28 to Day -1) and a Baseline Period (Day 1). During the Prerandomization Phase, participants will be divided into two cohorts based on the platelet count: Low Platelet Count Cohort and High Platelet Count Cohort. Participants in Low Platelet Count Cohort will be randomized to receive one of the four treatments: Placebo, Avatrombopag 20 mg, Avatrombopag 40 mg, or Avatrombopag 60 mg. Participants in High Platelet Count Cohort will be randomized to receive one of the three treatments: Placebo, Avatrombopag 20 mg, or Avatrombopag 40 mg.

The Randomization Phase includes the Treatment Period and the Follow-up Period. The Follow-up Period comprises 3 visits: Visit 4 (5 to 8 days after last dose of study drug [Study Day 10 to 13]), Visit 5 (12 to 15 days after last dose of study drug [Study Day 17 to 20]), and 30 days after receiving the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria

1. Japanese subjects greater than or equal to 20 years of age at Screening with chronic liver disease.
2. Subjects who have a mean baseline platelet count of less than 50 x 10^9/L. Platelet counts will be measured on 2 separate occasions, during the Screening Period and at Baseline, and must be performed at least one day apart with neither platelet count greater than 60 x 10^9/L.
3. Model For End-stage Liver Disease (MELD) score 24 at Screening.
4. If taking inhibitors of P glycoprotein (P-gp), except for verapamil, dose must be stable for 7 days prior to Screening.
5. Provide written informed consent.
6. Willing and able to comply with all aspects of the protocol.

Exclusion Criteria

1. Any history of arterial or venous thrombosis, including partial or complete thrombosis.
2. Evidence of thrombosis (partial or complete) in the main portal vein, portal vein branches, or any part of the splenic mesenteric system at Screening.
3. Portal vein blood flow velocity rate less than 10 cm/second at Screening.
4. Hepatic encephalopathy that cannot be effectively treated.
5. Subjects with HCC with Barcelona Clinic Liver Cancer (BCLC) staging classification C or D.
6. Platelet transfusion or receipt of blood products containing platelets within 7 days of Screening. However packed red blood cells are permitted.
7. Heparin, warfarin, nonsteroidal anti-inflammatory drugs (NSAID), aspirin, verapamil, and antiplatelet therapy with ticlopidine or glycoprotein IIb/IIIa antagonists (eg, tirofiban) within 7 days of Screening.
8. Use of erythropoietin stimulating agents within 7 days of Screening.
9. Interferon (IFN) use within 14 days of Screening.
10. Estrogen-containing hormonal contraceptive or hormone replacement therapy use within 30 days of Screening.
11. Active infection requiring systemic antibiotic therapy within 7 days of Screening. However, prophylactic use of antibiotics is permitted.
12. Alcohol abuse, alcohol dependence syndrome, drug abuse, or drug dependence within 6 months of the study start (unless participating in a controlled rehabilitation program) or acute alcoholic hepatitis (chronic alcoholic hepatitis is allowed) within 6 months of the study start.
13. Known to be human immunodeficiency virus positive.
14. Any clinically significant acute or active bleeding (eg, gastrointestinal, central nervous system).
15. Known history of any primary hematologic disorder (eg, immune thrombocytopenic purpura, myelodysplastic syndrome).
16. Known medical history of genetic prothrombotic syndromes (eg, Factor V Leiden; prothrombin G20210A; ATIII deficiency etc.)
17. Subjects with a history of significant cardiovascular disease (eg, congestive heart failure New York Heart Association Grade III/IV, arrhythmia known to increase the risk of thromboembolic events [eg, atrial fibrillation], coronary artery stent placement, angioplasty, and coronary artery bypass grafting).
18. Females of childbearing potential who have had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a progesterone only contraceptive implant/injection, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the subject must agree to use a double barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. All females will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months consecutive amenorrhea in the appropriate age group and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, hysterectomy, or bilateral oophorectomy) at least 1 month before dosing.
19. Females who are lactating or pregnant at Screening or Baseline (as documented by a positive serum beta-human chorionic gonadotropin [B-hCG] test with a minimum sensitivity 25 IU/L or equivalent units of B-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
20. Post liver transplant subjects.
21. Any subject who has previously received avatrombopag.
22. Hypersensitivity to avatrombopag maleate or any of its excipients.
23. Hemoglobin levels less than or equal to 8.0 or greater than or equal to 16.0 g/dL at Screening.
24. White blood cell count less than or equal to 1.5 x 10^9/L or greater than or equal to 15.0 x 10^9/L at Screening.
25. Serum sodium level less than or equal to 130 milliequivalents/L at Screening.
26. Current malignancy including solid tumors and hematologic malignancies (except HCC).
27. Any history of a medical condition or a concomitant medical condition that, in the opinion of the investigator(s), would compromise the subject's ability to safely complete the study.
28. Currently enrolled in another clinical trial or used any investigational drug or device within 30 days of Screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Japan (14):
  - Matsuyama, Ehime
  - Iizuka, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Kure, Hiroshima
  - Sapporo, Hokkaido
  - Sagamihara, Kanagawa
  - Ikeda, Osaka
  - Takatsuki, Osaka
  - Minato-Ku, Tokyo
  - Fukuoka
  - Kumamoto
  - Osaka
  - Yamanashi

REFERENCES:
- [Derived] Eguchi Y, Takahashi H, Mappa S, Santagostino E. Phase 2 study of avatrombopag in Japanese patients with chronic liver disease and thrombocytopenia. Hepatol Res. 2022 Apr;52(4):371-380. doi: 10.1111/hepr.13755. Epub 2022 Feb 21. PMID 35134259

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 56 participants were screened to enter into the study. Of these, 17 participants were screening failures, and 39 were randomized into the study. Of the 17 screening failures, 14 participants failed to meet the inclusion/exclusion criteria, 1 participant withdrew consent, and 2 participants were excluded for scheduling conflicts.
Groups:
- Placebo (60 mg): Participants took 60 milligrams (mg) placebo (3 x 20 mg matching placebo tablets) orally after a meal, once daily for 5 days.
- Avatrombopag (20 mg): Participants took 20 mg avatrombopag (1 x 20 mg avatrombopag tablet and 2 x 20 mg matching placebo tablets) orally after a meal, once daily for 5 days.
- Avatrombopag (40 mg): Participants took 40 mg avatrombopag (2 x 20 mg avatrombopag tablets and 1 x 20 mg matching placebo tablet) orally after a meal, once daily for 5 days.
- Avatrombopag (60 mg): Participants took 60 mg avatrombopag (3 x 20 mg avatrombopag tablets) orally, after a meal, once daily for 5 days.
Period: Overall Study
Arm/Group | Placebo (60 mg) | Avatrombopag (20 mg) | Avatrombopag (40 mg) | Avatrombopag (60 mg)
Started | 11 | 7 | 11 | 10
Completed | 11 | 7 | 11 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS was the group of randomized participants who received at least 1 dose of study drug.
Groups:
- Placebo (60 mg): Participants took 60 mg placebo (3 x 20 mg matching placebo tablets) orally after a meal, once daily for 5 days.
- Avatrombopag (40 mg): Avatrombopag (40 mg), Participants took 40 mg avatrombopag (2 x 20 mg avatrombopag tablets and 1 x 20 mg matching placebo tablet) orally after a meal, once daily for 5 days.
- Total: Total of all reporting groups
Arm/Group | Placebo (60 mg) | Avatrombopag (20 mg) | Avatrombopag (40 mg) | Avatrombopag (60 mg) | Total
Number analyzed (Participants) | 11 | 7 | 11 | 10 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (8.49) | 64.6 (8.42) | 64.6 (9.59) | 62.1 (7.32) | 65.8 (8.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5 | 3 | 13
  Male | 7 | 6 | 6 | 7 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Platelet Count Greater Than or Equal to 50 x 10^9/L and at Least 20 x 10^9/L Increase From Baseline at Visit 4
Description: Responders were defined as participants whose platelet count was greater than or equal to 50×10^9/liter (L) and change from baseline was at least 20×10^9/L at Visit 4. Participants receiving a platelet transfusion prior to the platelet count assessment at Visit 4 were considered as non-responders in the analysis. Two-sided 95% confidence interval (CI) is calculated by Clopper and Pearson method.
Time Frame: Baseline and Visit 4 (Day 10)
Population: Full Analysis Set (FAS) included all randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (60 mg) | Avatrombopag (20 mg) | Avatrombopag (40 mg) | Avatrombopag (60 mg)
Number analyzed (Participants) | 11 | 7 | 11 | 10
Percentage of participants | 9.1 [0.2 to 41.3] | 28.6 [3.7 to 71.0] | 63.6 [30.8 to 89.1] | 40.0 [12.2 to 73.8]
Statistical Analysis 1: Comparison: Placebo (60 mg) vs Avatrombopag (20 mg); Test type: Other; p = 0.146, Shirley-Williams test; P-value is based on Shirley-Williams test at a one-sided significance level of α = 0.025; Difference of responder rate vs. placebo = 19.5, 95% CI 2-sided [-18.1 to 57.0] — Difference of responder rate vs. placebo = responder rate for avatrombopag - responder rate for placebo; 95% CI is calculated based on normal approximation
Statistical Analysis 2: Comparison: Placebo (60 mg) vs Avatrombopag (40 mg); Test type: Other; p = 0.004, Shirley-Williams test; P-value is based on Shirley-Williams test at a one-sided significance level of α = 0.025; Difference of responder rate vs. placebo = 54.5, 95% CI 2-sided [21.4 to 87.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo (60 mg) vs Avatrombopag (60 mg); Test type: Other; p = 0.024, Shirley-Williams test; P-value is based on Shirley-Williams test at a one-sided significance level of α = 0.025; Difference of responder rate vs. placebo = 30.9, 95% CI 2-sided [-3.9 to 65.7] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Percentage of Participants With Platelet Count Greater Than or Equal to 50 x 10^9/L at Each Visit
Description: Responders were defined as the participants whose platelet count greater than or equal to 50 x 10^9/L by visit. Participants receiving a platelet transfusion prior to the platelet count assessment at Visit 4 were considered as non-responders in the analysis. Two-sided 95% CI is calculated by Clopper and Pearson method.
Time Frame: Visit 3 (Day 4 or 5), Visit 4 (Day 10), Visit 5 (Day 17) and Visit 6 (Day 35)
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (60 mg) | Avatrombopag (20 mg) | Avatrombopag (40 mg) | Avatrombopag (60 mg)
Number analyzed (Participants) | 11 | 7 | 11 | 10
Percentage of participants
  Visit 3 (Day 4 or Day 5) | 0.0 [0.0 to 28.5] | 14.3 [0.4 to 57.9] | 27.3 [6.0 to 61.0] | 0.0 [0.0 to 30.8]
  Visit 4 (Day 10) | 9.1 [0.2 to 41.3] | 71.4 [29.0 to 96.3] | 81.8 [48.2 to 97.7] | 50.0 [18.7 to 81.3]
  Visit 5 (Day 17) | 27.3 [6.0 to 61.0] | 0.0 [0.0 to 41.0] | 54.5 [23.4 to 83.3] | 20.0 [2.5 to 55.6]
  Visit 6 (Day 35) | 18.2 [2.3 to 51.8] | 0.0 [0.0 to 41.0] | 9.1 [0.2 to 41.3] | 0.0 [0.0 to 30.8]
Statistical Analysis 1: Comparison: Placebo (60 mg) vs Avatrombopag (20 mg); Visit 3 (Day 4 or Day 5); Test type: Other; p = 0.388, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α = 0.05; Difference of proportion vs. placebo = 14.3, 95% CI 2-sided [-11.6 to 40.2] — Difference of proportion vs. placebo = proportion of responders for avatrombopag - proportion of responders for placebo; 95% CI is calculated based on normal approximation
Statistical Analysis 2: Comparison: Placebo (60 mg) vs Avatrombopag (40 mg); Visit 3 (Day 4 or Day 5); Test type: Other; p = 0.214, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α = 0.05; Difference of proportion vs. placebo = 27.3, 95% CI 2-sided [1.0 to 53.6] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo (60 mg) vs Avatrombopag (20 mg); Visit 4 (Day 10); Test type: Other; p = 0.012, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α = 0.05; Difference of proportion vs. placebo = 62.3, 95% CI 2-sided [24.8 to 99.9] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Placebo (60 mg) vs Avatrombopag (40 mg); Visit 4 (Day 10); Test type: Other; p = 0.001, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α = 0.05; Difference of proportion vs. placebo = 72.7, 95% CI 2-sided [44.3 to 100.0] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo (60 mg) vs Avatrombopag (60 mg); Visit 4 (Day 10); Test type: Other; p = 0.063, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α = 0.05; Difference of proportion vs. placebo = 40.9, 95% CI 2-sided [5.6 to 76.2] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Placebo (60 mg) vs Avatrombopag (20 mg); Visit 5 (Day 17); Test type: Other; p = 0.245, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α = 0.05; Difference of proportion vs. placebo = -27.3, 95% CI 2-sided [-53.6 to -1.0] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Placebo (60 mg) vs Avatrombopag (40 mg); Visit 5 (Day 17); Test type: Other; p = 0.386, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α = 0.05; Difference of proportion vs. placebo = 27.3, 95% CI 2-sided [-12.2 to 66.8] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Placebo (60 mg) vs Avatrombopag (60 mg); Visit 5 (Day 17); Test type: Other; p = 1.000, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α = 0.05; Difference of proportion vs. placebo = -7.3, 95% CI 2-sided [-43.4 to 28.9] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Placebo (60 mg) vs Avatrombopag (20 mg); Visit 6 (Day 35); Test type: Other; p = 0.496, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α = 0.05; Difference of proportion vs. placebo = -18.2, 95% CI 2-sided [-41.0 to 4.6] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Placebo (60 mg) vs Avatrombopag (40 mg); Visit 6 (Day 35); Test type: Other; p = 1.000, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α = 0.05; Difference of proportion vs. placebo = -9.1, 95% CI 2-sided [-37.5 to 19.3] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: Placebo (60 mg) vs Avatrombopag (60 mg); Visit 6 (Day 35); Test type: Other; p = 0.476, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α = 0.05; Difference of proportion vs. placebo = -18.2, 95% CI 2-sided [-41.0 to 4.6] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percentage of Participants With Platelet Count Greater Than or Equal to 75 x 10^9/L at Each Visit
Description: Responders were defined as the participants whose platelet count greater than or equal to 75 x 10^9/L by visit. Participants receiving a platelet transfusion prior to the platelet count assessment at Visit 4 were considered as non-responders in the analysis. Two-sided 95% CI is calculated by Clopper and Pearson method.
Time Frame: Visit 3 (Day 4 or 5), Visit 4 (Day 10), Visit 5 (Day 17) and Visit 6 (Day 35)
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo (60 mg) | Avatrombopag (20 mg) | Avatrombopag (40 mg) | Avatrombopag (60 mg)
Number analyzed (Participants) | 11 | 7 | 11 | 10
Percentage of participants
  Visit 3 (Day 4 or Day 5) | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 30.8]
  Visit 4 (Day 10) | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 41.0] | 63.6 [30.8 to 89.1] | 30.0 [6.7 to 65.2]
  Visit 5 (Day 17) | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 28.5] | 10.0 [0.3 to 44.5]
  Visit 6 (Day 35) | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 41.0] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 30.8]
Statistical Analysis 1: Comparison: Placebo (60 mg) vs Avatrombopag (40 mg); Visit 4 (Day 10); Test type: Other; p = 0.003, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α= 0.05; Difference of proportion vs. placebo = 63.6, 95% CI 2-sided [35.2 to 92.1] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo (60 mg) vs Avatrombopag (60 mg); Visit 4 (Day 10); Test type: Other; p = 0.090, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α= 0.05; Difference of proportion vs. placebo = 30.0, 95% CI 2-sided [1.6 to 58.4] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo (60 mg) vs Avatrombopag (60 mg); Visit 5 (Day 17); Test type: Other; p = 0.476, Fisher Exact — P-value is based on Fisher's exact test at a two-sided significance level of α= 0.05; Difference of proportion vs. placebo = 10.0, 95% CI 2-sided [-8.6 to 28.6] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Percentage of Participants With Platelet Count Greater Than or Equal to 150 x 10^9/L At Each Visit
Description: Responders were defined as the participants whose platelet count greater than or equal to 150 x 10^9/L by visit. Participants receiving a platelet transfusion prior to the platelet count assessment at Visit 4 were considered as non-responders in the analysis.
Time Frame: Visit 3 (Day 4 or 5), Visit 4 (Day 10), Visit 5 (Day 17) and Visit 6 (Day 35)
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (60 mg) | Avatrombopag (20 mg) | Avatrombopag (40 mg) | Avatrombopag (60 mg)
Number analyzed (Participants) | 11 | 7 | 11 | 10
Percentage of participants
  Visit 3 (Day 4 or Day 5) | 0.0 | 0.0 | 0.0 | 0.0
  Visit 4 (Day 10) | 0.0 | 0.0 | 0.0 | 0.0
  Visit 5 (Day 17) | 0.0 | 0.0 | 0.0 | 0.0
  Visit 6 (Day 35) | 0.0 | 0.0 | 0.0 | 0.0

5. Secondary Outcome: Percentage of Participants With Platelet Count Greater Than or Equal to 200 x 10^9/L At Each Visit
Description: Responders were defined as the participants whose platelet count greater than or equal to 200 x 10^9/L by visit. Participants receiving a platelet transfusion prior to the platelet count assessment at Visit 4 were considered as non-responders in the analysis.
Time Frame: Visit 3 (Day 4 or 5), Visit 4 (Day 10), Visit 5 (Day 17) and Visit 6 (Day 35)
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (60 mg) | Avatrombopag (20 mg) | Avatrombopag (40 mg) | Avatrombopag (60 mg)
Number analyzed (Participants) | 11 | 7 | 11 | 10
Percentage of participants
  Visit 3 (Day 4 or Day 5) | 0.0 | 0.0 | 0.0 | 0.0
  Visit 4 (Day 10) | 0.0 | 0.0 | 0.0 | 0.0
  Visit 5 (Day 17) | 0.0 | 0.0 | 0.0 | 0.0
  Visit 6 (Day 35) | 0.0 | 0.0 | 0.0 | 0.0

6. Secondary Outcome: Platelet Count and Change From Baseline in Platelet Count by Visit
Time Frame: Baseline, Visit 3 (Day 4 or 5), Visit 4 (Day 10), Visit 5 (Day 17) and Visit 6 (Day 35)
Population: FAS
Measure: Mean (Standard Deviation); unit: Number of platelets x 10^9/L
Arm/Group | Placebo (60 mg) | Avatrombopag (20 mg) | Avatrombopag (40 mg) | Avatrombopag (60 mg)
Number analyzed (Participants) | 11 | 7 | 11 | 10
Number of platelets x 10^9/L
  Visit 2 (Baseline) Platelet count | 40.59 (7.024) | 40.57 (5.556) | 41.23 (5.159) | 28.85 (7.568)
  Visit 3 (Day 4 or Day 5) Platelet count | 41.27 (8.344) | 44.71 (6.102) | 46.09 (8.860) | 32.70 (9.967)
  Visit 3 (Day 4 or Day 5) Change from baseline | 0.68 (2.848) | 4.14 (7.099) | 4.86 (6.569) | 3.85 (6.223)
  Visit 4 (Day 10) Platelet count | 43.91 (10.568) | 53.29 (5.678) | 79.36 (24.800) | 55.90 (22.507)
  Visit 4 (Day 10) Change from baseline | 3.32 (7.163) | 12.71 (9.486) | 38.14 (22.781) | 27.05 (22.700)
  Visit 5 (Day 17) Platelet count | 40.10 (9.916) | 41.33 (4.803) | 55.73 (14.826) | 41.80 (16.578)
  Visit 5 (Day 17) Change from baseline: number analyzed (Participants) | 10 | 6 | 11 | 10
  Visit 5 (Day 17) Change from baseline | 0.40 (5.243) | 1.75 (3.402) | 14.50 (11.874) | 12.95 (12.857)
  Visit 6 (Day 35) Platelet count: number analyzed (Participants) | 10 | 6 | 11 | 9
  Visit 6 (Day 35) Platelet count | 41.50 (10.845) | 39.67 (5.574) | 41.36 (8.262) | 31.44 (8.353)
  Visit 6 (Day 35) Change from baseline: number analyzed (Participants) | 10 | 6 | 11 | 9
  Visit 6 (Day 35) Change from baseline | 1.80 (4.614) | 0.08 (1.686) | 0.14 (8.382) | 2.33 (4.265)
Statistical Analysis 1: Comparison: Placebo (60 mg) vs Avatrombopag (20 mg); Visit 3 (Day 4 or Day 5); Test type: Other; p = 0.296, Wilcoxon (Mann-Whitney) — P-value is based on Wilcoxon rank sum test at a two-sided significance level of α = 0.05 for each avatrombopag treatment group vs. placebo
Statistical Analysis 2: Comparison: Placebo (60 mg) vs Avatrombopag (40 mg); Visit 3 (Day 4 or Day 5); Test type: Other; p = 0.070, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 3: Comparison: Placebo (60 mg) vs Avatrombopag (60 mg); Visit 3 (Day 4 or Day 5); Test type: Other; p = 0.138, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 4: Comparison: Placebo (60 mg) vs Avatrombopag (20 mg); Visit 4 (Day 10); Test type: Other; p = 0.012, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 5: Comparison: Placebo (60 mg) vs Avatrombopag (40 mg); Visit 4 (Day 10); Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 6: Comparison: Placebo (60 mg) vs Avatrombopag (60 mg); Visit 4 (Day 10); Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 7: Comparison: Placebo (60 mg) vs Avatrombopag (20 mg); Visit 5 (Day 17); Test type: Other; p = 0.624, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 8: Comparison: Placebo (60 mg) vs Avatrombopag (40 mg); Visit 5 (Day 17); Test type: Other; p = 0.009, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 9: Comparison: Placebo (60 mg) vs Avatrombopag (60 mg); Visit 5 (Day 17); Test type: Other; p = 0.010, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 10: Comparison: Placebo (60 mg) vs Avatrombopag (20 mg); Visit 6 (Day 35); Test type: Other; p = 0.154, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 11: Comparison: Placebo (60 mg) vs Avatrombopag (40 mg); Visit 6 (Day 35); Test type: Other; p = 0.216, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 6, analysis 1]
Statistical Analysis 12: Comparison: Placebo (60 mg) vs Avatrombopag (60 mg); Visit 6 (Day 35); Test type: Other; p = 0.901, Wilcoxon (Mann-Whitney) — [p-value comment as in outcome 6, analysis 1]

7. Other Pre Specified Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Safety assessments consisted of monitoring and recording all AEs and SAEs, regular monitoring of hematology, blood chemistry, and urine values; periodic measurement of vital signs and electrocardiograms; physical examinations; and Doppler sonography. AE severity was graded using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, where Grade 1 = mild, Grade 2 = moderate, Grade 3 = Severe, Grade 4 = Life-threatening, and Grade 5 = Death related to the AE. All AEs graded as 4 or 5 were considered to be serious. A treatment-emergent adverse event (TEAE) was defined as an AE that started on or after the date of first dose of study drug, up to 30 days after the last dose of study drug. For each category, a participant with two or more adverse events in that category was counted only once. Treatment-related TEAEs were considered by the investigator to be possibly or probably related to study drug or TEAEs with a missing causality.
Time Frame: From the date of first dose of study drug up to 30 days after the last dose of the study drug, up to approximately 10 months
Population: Safety Analysis Set included all participants who received at least one dose of study drug and had at least one safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo (3 x 20 mg matching placebo tablets) received after a meal once daily for 5 days
- Avatrombopag 20-mg: 20 mg avatrombopag (1 x 20 mg tablet and 2 x 20 mg matching placebo tablets) received after a meal once daily for 5 days
- Avatrombopag 40-mg: 40 mg avatrombopag (2 x 20 mg tablets and 1 x 20 mg matching placebo tablet) received after a meal once daily for 5 days
- Avatrombopag 60-mg: 60 mg avatrombopag (3 x 20 mg tablets) received after a meal once daily for 5 days
Arm/Group | Placebo | Avatrombopag 20-mg | Avatrombopag 40-mg | Avatrombopag 60-mg
Number analyzed (Participants) | 11 | 7 | 11 | 10
Participants
  All TEAEs | 8 | 4 | 8 | 3
  Treatment-related TEAEs | 0 | 2 | 2 | 0
  Serious TEAEs | 0 | 0 | 0 | 0
  TEAEs leading to study drug dose adjustment | 0 | 0 | 0 | 0
  TEAEs leading to study drug withdrawal | 0 | 0 | 0 | 0
  TEAEs leading to study drug dose reduction | 0 | 0 | 0 | 0
  TEAEs leading to study drug dose interruption | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Number of Participants With Treatment-emergent Markedly Abnormal Laboratory Value (TEMAV) for Haematology
Time Frame: From the date of Screening until the date of last dose of study drug plus 30 days (Approximately 10 months)
Population: The safety analysis set was the group of participants who received at least 1 dose of study drug and had at least 1 postdose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avatrombopag 20-mg | Avatrombopag 40-mg | Avatrombopag 60-mg
Number analyzed (Participants) | 11 | 7 | 11 | 10
Participants
  Hemoglobin | 1 | 0 | 0 | 1
  Leukocytes | 4 | 4 | 2 | 0
  Alkaline phosphatase (ALP) | 1 | 0 | 0 | 0
  Alanine aminotransferase (ALT) | 0 | 0 | 0 | 1
  Bilirubin | 1 | 1 | 2 | 2
  Gamma-glutamyl transferase (γ-GTP) | 0 | 0 | 0 | 1
  Calcium | 0 | 0 | 0 | 2
  Albumin | 1 | 1 | 1 | 0
  Glucose | 3 | 2 | 2 | 1
  Triglycerides | 9 | 0 | 1 | 0
  Aspartate aminotransferase (AST) | 0 | 1 | 0 | 1

9. Other Pre Specified Outcome: Number of Participants With Clinically Significant Findings in Laboratory Values for Serum
Time Frame: From the date of Screening until the date of last dose of study drug plus 30 days (Approximately 10 months)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avatrombopag 20-mg | Avatrombopag 40-mg | Avatrombopag 60-mg
Number analyzed (Participants) | 11 | 7 | 11 | 10
Participants | 0 | 0 | 0 | 0

10. Other Pre Specified Outcome: Number of Participants With Clinically Significant Findings in Laboratory Values for Urinalysis
Time Frame: From the date of Screening until the date of last dose of study drug plus 30 days (Approximately 10 months)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avatrombopag 20-mg | Avatrombopag 40-mg | Avatrombopag 60-mg
Number analyzed (Participants) | 11 | 7 | 11 | 10
Participants | 0 | 0 | 0 | 0

11. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Sign Values
Time Frame: From the date of Screening until the date of last dose of study drug plus 30 days (Approximately 10 months)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avatrombopag 20-mg | Avatrombopag 40-mg | Avatrombopag 60-mg
Number analyzed (Participants) | 11 | 7 | 11 | 10
Participants | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Number of Participants With Markedly Abnormal Electrocardiographs
Time Frame: From the date of Screening until the date of last dose of study drug plus 30 days (Approximately 10 months)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Avatrombopag 20-mg | Avatrombopag 40-mg | Avatrombopag 60-mg
Number analyzed (Participants) | 11 | 7 | 11 | 10
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the date of first dose of study drug up to 30 days after the last dose of the study drug, up to approximately 10 months.
Description: Treatment-emergent adverse events and serious adverse events are reported. All adverse events were graded on a 5-point scale according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The safety analysis set was analyzed and included all participants who received at least one dose of study drug and had at least one post dose safety assessment. This set was analyzed "as treated."
Arm/Group | Placebo (60 mg) | Avatrombopag (20 mg) | Avatrombopag (40 mg) | Avatrombopag (60 mg)
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/7 | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/7 | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 8/11 | 4/7 | 8/11 | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (60 mg) (N=11) | Avatrombopag (20 mg) (N=7) | Avatrombopag (40 mg) (N=11) | Avatrombopag (60 mg) (N=10)
Conjunctival Haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Injection Site Reaction (General disorders) | 0 | 1 | 0 | 0
Puncture Site Pain (General disorders) | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 0 | 1 | 0
Vessel Puncture Site Haematoma (General disorders) | 0 | 1 | 0 | 0
Acute Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 1
Post Embolisation Syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0
Blood Glucose Increased (Investigations) | 1 | 1 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eczema Asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other